CLINICAL TRIAL: NCT03526861
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-centre Trial to Evaluate the Efficacy, Safety, and Tolerability of Tralokinumab Monotherapy in Adolescent Subjects With Moderate-to-severe Atopic Dermatitis (AD) Who Are Candidates for Systemic Therapy
Brief Title: Tralokinumab Monotherapy for Adolescent Subjects With Moderate to Severe Atopic Dermatitis - ECZTRA 6 (ECZema TRAlokinumab Trial no. 6).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0162-1334; 2017-005143-33 (EudraCT Number)
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Results first posted 2021-10-29 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-05

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Neither the subject nor any of the investigator or LEO staff who are involved in the treatment or clinical evaluation and monitoring of the subjects will be aware of the treatment received. The packaging and labelling of the investigational medicinal products (IMPs) will contain no evidence of their identity. Since tralokinumab and placebo are visually distinct and not matched for viscosity, IMP will be handled and administered by a qualified, unblinded healthcare professional at the site who will not be involved in the management of trial subjects and who will not perform any of the assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Tralokinumab(Dose1) initial-> Tralokinumab(Dose1) maintenanceA (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 1) loading SC injection on Day 0 followed by tralokinumab (Dose 1) injection regimen A.
  Week 16 to 52 (maintenance period):
  Tralokinumab (Dose 1) maintenance SC injection regimen A.
  Interventions: Drug: Tralokinumab
- Tralokinumab(Dose1) initial-> Tralokinumab(Dose1) maintenanceB (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 1) loading SC injection on Day 0 followed by tralokinumab (Dose 1) injection regimen A.
  Week 16 to 52 (maintenance period):
  Tralokinumab (Dose 1) maintenance SC injection regimen B.
  Interventions: Drug: Tralokinumab
- Tralokinumab(Dose2) initial-> Tralokinumab(Dose2) maintenanceA (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 2) loading SC injection on Day 0 followed by tralokinumab (Dose 2) injection regimen A.
  Week 16 to 52 (maintenance period):
  Tralokinumab (Dose 2) maintenance SC injection regimen A.
  Interventions: Drug: Tralokinumab
- Tralokinumab(Dose2) initial-> Tralokinumab(Dose2) maintenanceB (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 2) loading SC injection on Day 0 followed by tralokinumab (Dose 2) injection regimen A.
  Week 16 to 52 (maintenance period):
  Tralokinumab (Dose 2) maintenance SC injection regimen B.
  Interventions: Drug: Tralokinumab
- Placebo initial-> Placebo maintenance (Experimental): Week 0 to 16 (initial period):
  Placebo loading SC injection on Day 0 followed by placebo injection regimen A.
  Week 16 to 52 (maintenance period):
  Placebo continuation SC injection regimen A.
  Interventions: Drug: Placebos
- Tralokinumab (Dose1) initial-> Open-label tralokinumab (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 1) loading SC injection on Day 0 followed by tralokinumab (Dose 1) injection regimen A.
  Week 16 to 52:
  Tralokinumab (Dose 1) maintenance SC regimen A - open-label with allowed use of topical corticosteroids
  Interventions: Drug: Tralokinumab
- Tralokinumab (Dose2) initial-> Open-label tralokinumab (Experimental): Week 0 to 16 (initial period):
  Tralokinumab (Dose 2) loading SC injection on Day 0 followed by tralokinumab (Dose 2) injection regimen A.
  Week 16 to 52:
  Tralokinumab (Dose 1) maintenance SC regimen A - open-label with allowed use of topical corticosteroids
  Interventions: Drug: Tralokinumab
- Placebo initial-> Open-label tralokinumab (Experimental): Week 0 to 16 (initial period):
  Placebo loading SC injection on Day 0 followed by placebo injection regimen A.
  Week 16 to 52:
  Tralokinumab (Dose 1) maintenance SC regimen A - open-label with allowed use of topical corticosteroids
  Interventions: Drug: Tralokinumab; Drug: Placebos

INTERVENTIONS:
Drug: Tralokinumab — Tralokinumab is a human recombinant monoclonal antibody of the immunoglobulin G4 (IgG4) subclass that specifically binds to human interleukin (IL) 13 and blocks interaction with the IL-13 receptors.
  Arms: Placebo initial-> Open-label tralokinumab; Tralokinumab (Dose1) initial-> Open-label tralokinumab; Tralokinumab (Dose2) initial-> Open-label tralokinumab; Tralokinumab(Dose1) initial-> Tralokinumab(Dose1) maintenanceA; Tralokinumab(Dose1) initial-> Tralokinumab(Dose1) maintenanceB; Tralokinumab(Dose2) initial-> Tralokinumab(Dose2) maintenanceA; Tralokinumab(Dose2) initial-> Tralokinumab(Dose2) maintenanceB
Drug: Placebos — Placebo contains the same excipients in the same concentration only lacking tralokinumab.
  Other Names: Placebo
  Arms: Placebo initial-> Open-label tralokinumab; Placebo initial-> Placebo maintenance

SUMMARY:
Primary objective:

To evaluate the efficacy of subcutaneous (SC) administration of tralokinumab compared with placebo in treating adolescent subjects (age 12 to <18 years) with moderate-to-severe AD.

Secondary objectives:

To evaluate the efficacy of tralokinumab on severity and extent of AD, itch, and health-related quality of life compared with placebo.

To investigate the safety, immunogenicity, and tolerability of SC administration of tralokinumab compared with placebo when used to treat adolescent subjects (age 12 to <18 years) with moderate-to-severe AD.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 17.
* Diagnosis of AD as defined by the Hanifin and Rajka (1980) criteria for AD.
* History of AD for ≥1 year.
* History of topical corticosteroid (TCS; Europe: Class 3 or higher; US: Class 4 or lower) and/or topical calcineurin inhibitor (TCI) treatment failure or subjects for whom these topical AD treatments are medically inadvisable.
* AD involvement of ≥10% body surface area at screening and baseline.
* Stable dose of emollient twice daily (or more, as needed) for at least 14 days before randomisation.

Exclusion Criteria:

* Active dermatologic conditions that may confound the diagnosis of AD.
* Use of tanning beds or phototherapy within 6 weeks prior to randomisation.
* Treatment with systemic immunosuppressive/immunomodulating drugs and/or systemic corticosteroid within 4 weeks prior to randomisation.
* Treatment with TCS, TCI, or topical phosphodiesterase 4 (PDE-4) inhibitor within 2 weeks prior to randomisation.
* Receipt of any marketed biological therapy (i.e. immunoglobulin, anti immunoglobulin E) including dupilumab or investigational biologic agents.
* Active skin infection within 1 week prior to randomisation.
* Clinically significant infection within 4 weeks prior to randomisation.
* A helminth parasitic infection within 6 months prior to the date informed consent is obtained.
* Tuberculosis requiring treatment within the 12 months prior to screening.
* Known primary immunodeficiency disorder.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2021-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical expert, Study Director — LEO Pharma
Locations (76):
- United States (28):
  - LEO Pharma Investigational Site, Birmingham, Alabama
  - LEO Pharma Investigational Site, Fort Smith, Arkansas
  - Leo Pharma Investigational Site, Fountain Valley, California
  - LEO Pharma Investigational Site, Los Angeles, California
  - LEO Pharma Investigational Site, San Francisco, California
  - LEO Pharma Investigational Site, Stanford, California
  - LEO Pharma Investigational Site, New Haven, Connecticut
  - LEO Pharma Investigational Site, Miami, Florida
  - Leo Pharma Investigational Site, Albany, Georgia
  - LEO Pharma Investigational Site, Chicago, Illinois
  - LEO Pharma Investigational Site, Louisville, Kentucky
  - LEO Pharma Investigational Site, Baton Rouge, Louisiana
  - LEO Pharma Investigational Site, Ann Arbor, Michigan
  - LEO Pharma Investigational Site, Ypsilanti, Michigan
  - LEO Pharma Investigational Site, Minneapolis, Minnesota
  - LEO Pharma Investigational Site, East Windsor, New Jersey
  - LEO Pharma Investigational Site, Corning, New York
  - Leo Pharma Investigational Site, New York, New York
  - LEO Pharma Investigational Site, High Point, North Carolina
  - LEO Pharma Investigational Site, Bexley, Ohio
  - Leo Pharma Investigational Site, Tulsa, Oklahoma
  - LEO Pharma Investigational Site, Portland, Oregon
  - LEO Pharma Investigational Site, Philadelphia, Pennsylvania
  - Leo Pharma Investigational Site, North Charleston, South Carolina
  - Leo Pharma Investigational Site, Murfreesboro, Tennessee
  - LEO Pharma Investigational Site, Austin, Texas
  - LEO Pharma Investigational Site, Houston, Texas
  - Leo Pharma Investigational Site, San Antonio, Texas
- Australia (4):
  - Leo Pharma Investigationel Site, Darlinghurst
  - Leo Pharma Investigationel Site, Kogarah
  - Leo Pharma Investigationel Site, Melbourne
  - Leo Pharma Investigationel Site, Woolloongabba
- Belgium (4):
  - Leo Pharma Investigationel Site, Brussels
  - Leo Pharma Investigationel Site, Ghent
  - Leo Pharma Investigationel Site, Liège
  - Leo Pharma Investigational Site, Maldegem
- Canada (10):
  - LEO Pharma Investigational Site, Calgary, Alberta
  - LEO Pharma Investigational Site, Edmonton, Alberta
  - LEO Pharma Investigational Site, Surrey, British Columbia
  - LEO Pharma Investigational Site, Winnipeg, Manitoba
  - LEO Pharma Investigational Site, Markham, Ontario
  - LEO Pharma Investigational Site, Oakville, Ontario
  - LEO Pharma Investigational Site, Toronto, Ontario
  - LEO Pharma Investigational Site, Windsor, Ontario
  - LEO Pharma Investigational Site, Montreal, Quebec
  - LEO Pharma Investigational Site, Saskatoon, Saskatchewan
- France (4):
  - Leo Pharma Investigationel Site, Marseille
  - Leo Pharma Investigationel Site, Nice
  - Leo Pharma Investigationel Site, Paris
  - Leo Pharma Investigationel Site, Valence
- Germany (4):
  - Leo Pharma Investigationel Site, Berlin
  - Leo Pharma Investigationel Site, Dresden
  - Leo Pharma Investigationel Site, Jena
  - Leo Pharma Investigationel Site, Osnabrück
- Japan (11):
  - Leo Pharma Investigationel Site, Fukuoka
  - Leo Pharma Investigationel Site, Kagoshima
  - Leo Pharma Investigationel Site, Kyoto
  - Leo Pharma Investigationel Site, Nagoya
  - Leo Pharma Investigationel Site, Obihiro
  - Leo Pharma Investigationel Site, Osaka
  - Leo Pharma Investigationel Site, Osaka-fu
  - Leo Pharma Investigationel Site, Shimotsuke
  - Leo Pharma Investigationel Site, Tokyo
  - Leo Pharma Investigationel Site, Tsu
  - Leo Pharma Investigationel Site, Yamanashi
- Netherlands (4):
  - Leo Pharma Investigationel Site, Bergen op Zoom
  - Leo Pharma Investigationel Site, Breda
  - Leo Pharma Investigationel Site, Groningen
  - Leo Pharma Investigationel Site, Rotterdam
- Poland (5):
  - Leo Pharma Investigationel Site, Krakow
  - Leo Pharma Investigationel Site, Lodz
  - Leo Pharma Investigationel Site, Rzeszów
  - Leo Pharma Investigationel Site, Świdnik
  - Leo Pharma Investigationel Site, Wroclaw
- United Kingdom (2):
  - Leo Pharma Investigationel Site, Glasgow
  - Leo Pharma Investigationel Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Paller AS, Flohr C, Cork M, Bewley A, Blauvelt A, Hong HC, Imafuku S, Schuttelaar MLA, Simpson EL, Soong W, Arlert P, Lophaven KW, Kurbasic A, Soldbro L, Vest NS, Wollenberg A. Efficacy and Safety of Tralokinumab in Adolescents With Moderate to Severe Atopic Dermatitis: The Phase 3 ECZTRA 6 Randomized Clinical Trial. JAMA Dermatol. 2023 Jun 1;159(6):596-605. doi: 10.1001/jamadermatol.2023.0627. PMID 37074705
- [Derived] Paller AS, Blauvelt A, Soong W, Chih-Ho Hong H, Schuttelaar MLA, Schneider SKR, Simpson EL. Clinically Meaningful Improvements in Adolescents with Moderate-to-Severe Atopic Dermatitis Treated with Tralokinumab who did not Achieve Clear or Almost Clear Skin at Week 16. Dermatol Ther (Heidelb). 2025 Oct;15(10):2879-2896. doi: 10.1007/s13555-025-01484-1. Epub 2025 Jul 28. PMID 40721559
- [Derived] Paller AS, Soong W, Boguniewicz M, Geng B, Thyssen JP, Bennike N, Schneider S, Wollenberg A. Effect of tralokinumab on moderate-to-severe atopic dermatitis in patients with atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Oct;135(4):425-433.e4. doi: 10.1016/j.anai.2025.06.022. Epub 2025 Jun 22. PMID 40555305
- [Derived] Soehoel A, Larsen MS, Timmermann S. Population Pharmacokinetics of Tralokinumab in Adult Subjects With Moderate to Severe Atopic Dermatitis. Clin Pharmacol Drug Dev. 2022 Aug;11(8):910-921. doi: 10.1002/cpdd.1113. Epub 2022 Jun 7. PMID 35671038

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Treatment Period - Tralokinumab 300 mg Q2W: Week 0 to Week 16:
  Tralokinumab 300 mg Q2W Tralokinumab: Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for SC administration.
  At Day 0, each subject received 4 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab. At subsequent visits (Q2W) each subject received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Initial Treatment Period - Tralokinumab 150 mg Q2W: Week 0 to Week 16:
  Tralokinumab 150 mg Q2W. Tralokinumab: Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for SC administration.
  At Day 0, each subject received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab and 2 subcutaneous injections (each 1.0 mL) of placebo to receive a total loading dose of 300 mg tralokinumab. At subsequent visits (Q2W) each subject received 1 subcutaneous injection (1.0 mL) of 150 mg tralokinumab and 1 subcutaneous injection (1.0 mL) of placebo to receive a total dose of 150 mg tralokinumab.
- Initial Treatment Period - Placebo: Week 0 to Week 16:
  Placebo Q2W Placebo: Placebo contains the same excipients, in the same concentration, only lacking tralokinumab.
  At Day 0, each subject received 4 subcutaneous injections (each 1.0 mL) of placebo. At subsequent visits (Q2W) each subject received 2 subcutaneous injections (each 1.0 mL) of placebo.
- Maintenance Treatment Period - Tralokinumab 300 mg Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 and initially randomised to tralokinumab 300 mg Q2W, re-randomised to tralokinumab 300 mg Q2W maintenance dosing regimen. At each visit (Q2W), subject received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Maintenance Treatment Period - Tralokinumab 300 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 and initially randomised to tralokinumab 300 mg Q2W, re-randomised to tralokinumab 300 mg Q4W maintenance dosing regimen. At each visit (Q2W), subject received alternating dose administrations: 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab; or 2 subcutaneous injections (each 1.0 mL) of placebo.
- Maintenance Treatment Period - Tralokinumab 150 mg Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 and initially randomised to tralokinumab 150 mg Q2W, re-randomised to tralokinumab 150 mg Q2W maintenance dosing regimen. At each visit (Q2W), subject received 1 subcutaneous injection (1.0 mL) of 150 mg tralokinumab and 1 subcutaneous injection (1.0 mL) of placebo to receive a total dose of 150 mg tralokinumab.
- Maintenance Treatment Period - Tralokinumab 150 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 from Week 2 to Week 16 and initially randomised to tralokinumab 150 mg Q2W, re-randomised to tralokinumab 150 mg Q4W maintenance dosing regimen. At each visit (Q2W), subject received alternating dose administrations: 1 subcutaneous injection (1.0 mL) of 150 mg tralokinumab and 1 subcutaneous injection (1.0 mL) of placebo to receive a total dose of 150 mg tralokinumab; or 2 subcutaneous injections (each 1.0 mL) of placebo.
- Maintenance Treatment Period - Placebo Q2W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 and initially randomised to placebo, assigned to continue to placebo Q2W. At each visit (Q2W), subject received 2 subcutaneous injections (each 1.0 mL) of placebo.
- Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS: Week 16 to Week 52:
  Subjects receiving initial treatment with tralokinumab 150 mg/tralokinumab 300 mg/placebo Q2W who did not achieve clinical response at Week 16 without use of rescue medication from Week 2 to Week 16, assigned to open-label treatment at Week 16 with tralokinumab 300 mg Q2W regimen + optional topical corticosteroids (TCS) OR Subjects receiving maintenance treatment with tralokinumab 150 mg Q2W/Q4W, tralokinumab 300 mg Q2W/Q4W, or placebo Q2W assigned to open-label treatment after Week 16 with tralokinumab 300 mg Q2W regimen + optional TCS if
  * IGA of at least 2 and not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA=0 at Week 16.
  * IGA of at least 3 and not achieving EASI75 over at least a 4-week period (i.e. over 3 consecutive visits) for subjects with IGA=1 at Week 16.
  * Not achieving EASI75 over at least a 4-week period (over 3 consecutive visits) for subjects with IGA>1 at Week 16. At each visit, subjects received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab Q2W to receive a total dose of 300 mg.
Period: Initial Treatment Period
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS
Started | 101 | 100 | 100 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 94 | 93 | 86 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 7 | 14 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not dosed | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomised at site with quality/GCP issues identified, subject withdrawn from the trial | 3 | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject discontinued IMP before Week 16 | 3 | 5 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Treatment Period
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS
Started (Maintenance treatment period was in parallel to the open-label treatment period.) | 0 | 0 | 0 | 13 | 14 | 12 | 14 | 6 | 0
Completed | 0 | 0 | 0 | 5 | 8 | 8 | 8 | 4 | 0
Not Completed | 0 | 0 | 0 | 8 | 6 | 4 | 6 | 2 | 0
Not completed — Subject discontinued IMP between Week 16 and Week 52 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Not completed — Subject transferred to open-label treatment | 0 | 0 | 0 | 6 | 5 | 4 | 5 | 2 | 0
Not completed — Randomised at site with quality/GCP issues identified, subject withdrawn from the trial | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open-label Treatment Period
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W | Maintenance Treatment Period - Placebo Q2W | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS
Started (Open-label treatment period was in parallel to the maintenance treatment period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 242 (226 subjects transferred to open-label treatment at Week 16. 24 subjects transferred to open-label treatment between Week 16 and Week 52.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 214
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 28
Not completed — Subject discontinued IMP between Week 16 and Week 52 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19
Not completed — Completed treatment (received the last planned dose of IMP) and withdrew from the trial at Week 50 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Randomised at site with quality/GCP issues identified, subject withdrawn from the trial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Initial Treatment Period - Tralokinumab 300 mg Q2W: Week 0 to Week 16:
  Tralokinumab 300 mg Q2W Tralokinumab: Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration.
  At Day 0, each subject received 4 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total loading dose of 600 mg tralokinumab. At subsequent visits (Q2W) each subject received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab.
- Initial Treatment Period - Tralokinumab 150 mg Q2W: Week 0 to Week 16:
  Tralokinumab 150 mg Q2W. Tralokinumab: Tralokinumab is a human recombinant monoclonal antibody of the IgG4 subclass that specifically binds to human IL-13 and blocks interaction with the IL-13 receptors. It is presented as a liquid formulation for subcutaneous administration.
  At Day 0, each subject received 2 subcutaneous injections (each 1.0 mL) of 150 mg tralokinumab and 2 subcutaneous injections (each 1.0 mL) of placebo to receive a total loading dose of 300 mg tralokinumab. At subsequent visits (Q2W) each subject received 1 subcutaneous injection (1.0 mL) of 150 mg tralokinumab and 1 subcutaneous injection (1.0 mL) of placebo to receive a total dose of 150 mg tralokinumab.
- Total: Total of all reporting groups
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo | Total
Number analyzed (Participants) | 101 | 100 | 100 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.6 (1.8) | 14.8 (1.7) | 14.4 (1.6) | 14.6 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 46 | 146
  Male | 49 | 52 | 54 | 155
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 10 | 32
  Not Hispanic or Latino | 89 | 90 | 90 | 269
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59 | 56 | 58 | 173
  Black or African American | 14 | 8 | 12 | 34
  Asian | 21 | 28 | 23 | 72
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 4
  Other | 5 | 6 | 4 | 15
Region of Enrollment [Number; unit: participants]
  Canada | 21 | 19 | 12 | 52
  Netherlands | 4 | 4 | 5 | 13
  Belgium | 2 | 3 | 3 | 8
  United States | 31 | 33 | 41 | 105
  Japan | 11 | 10 | 11 | 32
  Poland | 19 | 20 | 15 | 54
  United Kingdom | 1 | 0 | 3 | 4
  Australia | 5 | 5 | 4 | 14
  France | 2 | 2 | 4 | 8
  Germany | 5 | 4 | 2 | 11
Investigator's Global Assessment [Count of Participants; unit: Participants] — The Investigator's Global Assessment (IGA) is an instrument used in clinical trials to rate the severity of the subject's global atopic dermatitis and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
  Participants
    Clear | 0 | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0 | 0
    Mild | 0 | 0 | 0 | 0
    Moderate | 52 | 55 | 54 | 161
    Severe | 48 | 44 | 45 | 137
    Missing | 1 | 1 | 1 | 3
Eczema Area and Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Eczema Area and Severity Index (EASI) is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
  units on a scale | 31.90 (13.74) | 31.89 (12.97) | 31.25 (14.19) | 31.68 (13.60)
Scoring Atopic Dermatitis [Mean (Standard Deviation); unit: units on a scale] — The Scoring Atopic Dermatitis (SCORAD) is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
  units on a scale | 68.41 (13.51) | 67.42 (14.51) | 67.70 (14.77) | 67.84 (14.23)
Children's Dermatology Life Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Children's Dermatology Life Quality Index (DLQI) consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life (QoL) over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). The total score is the sum of the 10 items (0 to 30); a high score is indicative of a poor health-related quality of life.
  units on a scale | 13.29 (7.18) | 12.86 (6.27) | 13.14 (5.99) | 13.10 (6.48)
Adolescent Worst Pruritus NRS (weekly average) [Mean (Standard Deviation); unit: units on a scale] — Subjects assessed their worst itch severity over the past 24 hours using an 11-point numeric rating scale ('Adolescent Worst Pruritus NRS') each morning, with 0 indicating 'no itch' and 10 indicating 'worst itch possible'.
  units on a scale | 7.79 (1.53) | 7.49 (1.58) | 7.45 (1.62) | 7.58 (1.58)
Body surface area affected by atopic dermatitis (AD) [Mean (Standard Deviation); unit: percentage affected] | 49.8 (23.0) | 52.0 (22.5) | 50.9 (23.5) | 50.9 (23.0)
Age of onset of atopic dermatitis (AD) [Mean (Standard Deviation); unit: years] | 2.5 (3.5) | 2.1 (3.3) | 2.4 (3.5) | 2.4 (3.4)
Duration of atopic dermatitis (AD) [Mean (Standard Deviation); unit: years] | 12.1 (3.7) | 12.7 (3.7) | 12.0 (3.4) | 12.3 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16
Description: The IGA is an instrument used in clinical trials to rate the severity of the subject's global AD and is based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Time Frame: At Week 16
Population: The full analysis set (FAS: All subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified) was used for the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 17 | 21 | 4
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects with IGA score of 0 (clear) or 1 (almost clear) at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoint tested sequentially at a 5% significance level; p = 0.002, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 13.8, 95% CI 2-sided [5.3 to 22.3] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects with IGA score of 0 (clear) or 1 (almost clear) at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoint tested sequentially at a 5% significance level; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 17.5, 95% CI 2-sided [8.4 to 26.6] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

2. Primary Outcome: Subjects With at Least 75% Reduction in Eczema Area and Severity Index (EASI75) at Week 16
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and/or more extensive condition.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 27 | 28 | 6
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 75% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoint tested sequentially at a 5% significance level; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 22.0, 95% CI 2-sided [12.0 to 32.0] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 75% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Primary endpoint tested sequentially at a 5% significance level; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 22.5, 95% CI 2-sided [12.4 to 32.6] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

3. Secondary Outcome: Subjects With Reduction of Adolescent Worst Pruritus Numeric Rating Scale (NRS) (Weekly Average) of at Least 4 From Baseline to Week 16
Description: The Adolescent Worst Pruritus NRS is used by subjects to assess their worst itch over the past 24 hours using an 11-point NRS with 0 indicating 'no itch' and 10 indicating 'worst itch possible'.
Time Frame: At Week 16
Population: Subjects in the full analysis set with baseline Adolescent Worst Pruritus weekly average ≥4. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 96 | 95 | 90
Participants | 24 | 22 | 3
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects with at least 4-point reduction in Adolescent Worst Pruritus NRS were considered responders. Subjects with missing data or who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Secondary endpoint tested sequentially at a 2.5% significance level; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 21.7, 95% CI 2-sided [12.3 to 31.1] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects with at least 4-point reduction in Adolescent Worst Pruritus NRS were considered responders. Subjects with missing data or who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — Secondary endpoint tested sequentially at a 5% significance level; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 19.9, 95% CI 2-sided [10.6 to 29.2] — Mantel-Haenszel risk difference, stratified by region and baseline disease severity

4. Secondary Outcome: Change in Scoring Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: The SCORAD is a validated tool to evaluate the extent and severity of AD lesions, along with subjective symptoms. The maximum total score is 103, with higher values indicating more severe disease.
Time Frame: From Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
units on a scale | -29.1 (2.4) | -27.5 (2.4) | -9.5 (3.0)
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Repeated measurements model on post-baseline data. In case of no post-baseline assessments before initiation of rescue medication, the Week 2 change was imputed as 0. Data collected after permanent discontinuation of IMP or after use of rescue treatment from Week 2 to Week 16 were not included in the analysis; Test type: Superiority — This secondary endpoint was tested sequentially using the Holm-Bonferroni method for multiplicity adjustment at a 2.5% significance level after the sequential testing of the primary endpoints and first secondary endpoint, if these showed statistical significance; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -19.7, 95% CI 2-sided [-27.1 to -12.2]
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — This secondary endpoint was tested sequentially using the Holm-Bonferroni method for multiplicity adjustment at a 5% significance level after the sequential testing of the primary endpoints and first secondary endpoint, if these showed statistical significance; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -18.0, 95% CI 2-sided [-25.6 to -10.4]

5. Secondary Outcome: Change in Children's Dermatology Life Quality Index (CDLQI) Score From Baseline to Week 16
Description: The CDLQI is a validated questionnaire with content specific to those with dermatology conditions. It consists of 10 items addressing the subject's perception of the impact of their skin disease on various aspects of their quality of life over the last week such as dermatology-related symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and the treatment. Each item is scored on a 4-point Likert scale (0 = 'not at all'; 1 = 'only a little'; 2 = 'quite a lot'; 3 = 'very much'). Item 7 (on school time) has one additional response category 'prevented school', which is also scored '3'. The total score of the CDLQI is the sum of the 10 items (0 to 30); a high score is indicative of a poor quality of life.
Time Frame: From Week 0 to Week 16
Population: Subjects in the full analysis set with non-missing baseline CDLQI score. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 94 | 95 | 89
units on a scale | -6.7 (0.6) | -6.1 (0.6) | -4.1 (0.7)
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.007, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -2.6, 95% CI 2-sided [-4.5 to -0.7]
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — [test comment as in outcome 4, analysis 2]; p = 0.040, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -2.0, 95% CI 2-sided [-3.9 to -0.1]

6. Secondary Outcome: Number of Adverse Events
Description: Number of AEs during the Initial treatment period is presented. For a summary of AEs and SAEs by MedDRA system organ class (SOC) and preferred term (PT) during the initial treatment period, maintenance treatment period, open-label treatment period, and safety follow-up period, see the Adverse Events Overview section.
Time Frame: From Week 0 to Week 16
Population: The analysis was performed on the safety analysis set. The safety analysis set comprised all subjects randomised to initial treatment and exposed to IMP, except for subjects randomised at the investigational sites where substantial quality/GCP issues were identified . The safety analysis set was identical to the full analysis set.
Measure: Number; unit: number of adverse events
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
number of adverse events | 130 | 175 | 134

7. Secondary Outcome: Presence of Anti-drug Antibodies
Description: Anti-tralokinumab antibody levels were analysed using a validated bioanalytical method.
Time Frame: From Week 0 to Week 16
Population: The analysis was performed on the safety analysis set. The safety analysis set comprised all subjects randomised to initial treatment, except for subjects randomised at the investigational sites where substantial quality/GCP issues were identified and subjects for whom no post-baseline safety data were available. The safety analysis set was identical to the full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 1 | 7 | 2

8. Secondary Outcome: Subjects With at Least 50% Reduction in Eczema Area and Severity Index (EASI50) at Week 16.
Description: as for outcome 2
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 50 | 45 | 13
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 50% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 38.5, 95% CI 2-sided [26.8 to 50.2] — Mantel-Haenszel risk difference, stratified by region and disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 50% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 32.4, 95% CI 2-sided [20.6 to 44.1] — Mantel-Haenszel risk difference, stratified by region and disease severity

9. Secondary Outcome: Subjects With at Least 90% Reduction in Eczema Area and Severity Index (EASI90) at Week 16.
Description: as for outcome 2
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 17 | 19 | 4
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 90% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p = 0.002, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 13.7, 95% CI 2-sided [5.2 to 22.2] — Mantel-Haenszel risk difference, stratified by region and disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 90% reduction in EASI at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 15.3, 95% CI 2-sided [6.5 to 24.1] — Mantel-Haenszel risk difference, stratified by region and disease severity

10. Secondary Outcome: Change in Eczema Area and Severity Index (EASI) Score From Baseline to Week 16
Description: as for outcome 2
Time Frame: From Week 0 to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
units on a scale | -18.1 (1.3) | -18.1 (1.4) | -8.7 (1.6)
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -9.4, 95% CI 2-sided [-13.5 to -5.3]
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -9.4, 95% CI 2-sided [-13.6 to -5.3]

11. Secondary Outcome: Subjects With at Least 75% Reduction in Scoring Atopic Dermatitis (SCORAD75) at Week 16
Description: The SCORAD is a validated tool to evaluate the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with a higher values indicating a more extensive and/or severe condition.
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 12 | 16 | 1
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 75% reduction in SCORAD at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p = 0.002, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 11.5, 95% CI 2-sided [4.5 to 18.4] — Mantel-Haenszel risk difference, stratified by region and disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 75% reduction in SCORAD at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 15.6, 95% CI 2-sided [7.8 to 23.3] — Mantel-Haenszel risk difference, stratified by region and disease severity

12. Secondary Outcome: Subjects With at Least 50% Reduction in Scoring Atopic Dermatitis (SCORAD50) at Week 16
Description: as for outcome 11
Time Frame: At Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 97 | 98 | 94
Participants | 30 | 30 | 5
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 50% reduction in SCORAD at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 26.2, 95% CI 2-sided [16.1 to 36.3] — Mantel-Haenszel risk difference, stratified by region and disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects who achieved at least 50% reduction in SCORAD at Week 16 were considered responders. Subjects with missing data or subjects who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 25.5, 95% CI 2-sided [15.3 to 35.7] — Mantel-Haenszel risk difference, stratified by region and disease severity

13. Secondary Outcome: Change in Adolescent Worst Pruritus Numeric Rating Scale (NRS) (Weekly Average) From Baseline to Week 16
Description: as for outcome 3
Time Frame: From Week 0 to Week 16
Population: Subjects in the full analysis set with non-missing baseline Adolescent Worst Pruritus NRS score. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 96 | 96 | 92
units on a scale | -3.0 (0.3) | -2.7 (0.3) | -1.5 (0.3)
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -1.5, 95% CI 2-sided [-2.4 to -0.6]
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p = 0.007, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -1.2, 95% CI 2-sided [-2.1 to -0.3]

14. Secondary Outcome: Participants With Reduction of Adolescent Worst Pruritus Numeric Rating Scale (NRS) (Weekly Average) of at Least 3 From Baseline to Week 16
Description: as for outcome 3
Time Frame: At Week 16
Population: Subjects in the full analysis set with baseline Adolescent Worst Pruritus weekly average ≥3. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 96 | 95 | 91
Participants | 28 | 29 | 8
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; Subjects with at least 3-point reduction in Adolescent Worst Pruritus NRS were considered responders. Subjects with missing data or who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 300 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 20.3, 95% CI 2-sided [9.7 to 31.0] — Mantel-Haenszel risk difference, stratified by region and disease severity
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; Subjects with at least 3-point reduction in Adolescent Worst Pruritus NRS were considered responders. Subjects with missing data or who received rescue medication from Week 2 to Week 16 were considered non-responders. Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity. The null hypothesis of no difference in response rate between tralokinumab 150 mg Q2W and placebo was tested against the 2-sided alternative that there is a difference; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Cochran-Mantel-Haenszel — Based on the primary analysis of the primary estimand 'composite'; Risk Difference (RD) = 21.8, 95% CI 2-sided [10.9 to 32.7] — Mantel-Haenszel risk difference, stratified by region and disease severity

15. Secondary Outcome: Change in Patient Oriented Eczema Measure (POEM) From Baseline to Week 16
Description: The POEM is a validated questionnaire used to assess disease symptoms in atopic eczema patients in both clinical practice and clinical trials. The tool consists of 7 items each addressing a specific symptom (itching, sleep, bleeding, weeping, cracking, flaking, and dryness). Subjects will score how often they have experienced each symptom over the previous week on a 5-point categorical response scale (0 = 'no days'; 1 = '1 to 2 days'; 2 = '3 to 4 days'; 3 = '5 to 6' days; 4 = 'every day'). The total score is the sum of the 7 items (range 0 to 28) and reflects disease-related morbidity; a high score is indicative of a worse disease severity.
Time Frame: From Week 0 to Week 16
Population: Subjects in the full analysis set with non-missing baseline POEM score. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W | Initial Treatment Period - Placebo
Number analyzed (Participants) | 94 | 95 | 87
units on a scale | -8.4 (0.8) | -7.8 (0.8) | -2.4 (1.0)
Statistical Analysis 1: Comparison: Initial Treatment Period - Tralokinumab 300 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -6.0, 95% CI 2-sided [-8.4 to -3.6]
Statistical Analysis 2: Comparison: Initial Treatment Period - Tralokinumab 150 mg Q2W vs Initial Treatment Period - Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — The statistical test was not controlled for multiplicity; p < 0.001, Repeated measurements model — Based on the primary analysis of the primary estimand 'hypothetical'; Difference of least square means = -5.4, 95% CI 2-sided [-7.9 to -3.0]

16. Secondary Outcome: Tralokinumab Serum Trough Concentration at Week 16
Description: Serum samples for determination of tralokinumab concentrations were analysed by a laboratory using a validated bioanalytical method.
Time Frame: At Week 16
Population: Subjects in the full analysis set who were randomised to tralokinumab. The full analysis set (FAS) comprised all subjects randomised to initial treatment who were exposed to IMP and not randomised at the investigational sites where substantial quality/GCP issues were identified.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Initial Treatment Period - Tralokinumab 300 mg Q2W | Initial Treatment Period - Tralokinumab 150 mg Q2W
Number analyzed (Participants) | 97 | 98
microgram/mL | 105.7 (39.0) | 56.4 (35.4)

17. Secondary Outcome: Subjects With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 52 Among Subjects With IGA Score of 0 or 1 at Week 16 After Initial Randomisation to Tralokinumab and Without Use of Rescue From Week 2 to Week 16
Description: as for outcome 1
Time Frame: At Week 52
Population: Subjects in the full analysis set (FAS) who were re-randomised to maintenance treatment and achieved an Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16 without use of rescue medication from Week 2 to Week 16.
Measure: Count of Participants; unit: Participants
Groups:
- Maintenance Treatment Period - Tralokinumab 300 mg Q4W: Week 16 to Week 52:
  Subjects achieving a clinical response at Week 16 without use of rescue medication from Week 2 to Week 16 and initially randomised to tralokinumab 300 mg Q2W, re-randomised to tralokinumab 300 mg Q4W maintenance dosing regimen. At each visit (Q2W), subject received alternating dose administrations: 2 subcutaneous injection (each 1.0 mL) of 150 mg tralokinumab to receive a total dose of 300 mg tralokinumab; or 2 subcutaneous injections (each 1.0 mL) of placebo.
Arm/Group | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W
Number analyzed (Participants) | 8 | 8 | 9 | 10
Participants | 3 | 7 | 6 | 6

18. Secondary Outcome: Subjects With at Least 75% Reduction in Eczema Area and Severity Index (EASI75) at Week 52 Among Subjects With at Least 75% Reduction in EASI at Week 16 After Initial Randomisation to Tralokinumab and Without Use of Rescue From Week 2 to Week 16
Description: as for outcome 2
Time Frame: At Week 52
Population: Subjects in the full analysis set (FAS) who were re-randomised to maintenance treatment and achieved at Least 75% Reduction in Eczema Area and Severity Index (EASI75) at Week 16 without use of rescue medication from Week 2 to Week 16.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W
Number analyzed (Participants) | 9 | 13 | 11 | 14
Participants | 4 | 7 | 7 | 7

19. Secondary Outcome: Tralokinumab Serum Trough Concentration at Week 66
Description: as for outcome 16
Time Frame: At Week 66
Population: 13 subjects in maintenance safety analysis set who were initially randomised to tralokinumab and completed the maintenance treatment period on treatment. 234 subjects in the open-label safety analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/mL
Arm/Group | Maintenance Treatment Period - Tralokinumab 300 mg Q2W | Maintenance Treatment Period - Tralokinumab 300 mg Q4W | Maintenance Treatment Period - Tralokinumab 150 mg Q2W | Maintenance Treatment Period - Tralokinumab 150 mg Q4W | Open-label Treatment -Tralokinumab 300 mg Q2W + Optional TCS
Number analyzed (Participants) | 1 | 5 | 4 | 3 | 234
microgram/mL | 5.9 (NA) — 1 subject provided data at Week 66, hence coefficient of variation could not be calculated. | 1.0 (458.0) | 1.5 (168.6) | 2.6 (75.6) | 4.4 (136.5)

ADVERSE EVENTS:
Time Frame: Initial Treatment Period: Week 0 to Week 16, Maintenance Treatment Period: Week 16 to Week 52, Open-label Treatment: Week 16 to Week 52; Safety Follow-up Period: Week 52 to Week 66.
Groups:
- Initial Treatment Period - Tralokinumab 300 Q2W: Initial Treatment Period - Tralokinumab 300 Q2W (n=97, PYE=29.48)
- Initial Treatment Period - Tralokinumab 150 Q2W: Initial Treatment Period - Tralokinumab 150 Q2W (n=98, PYE=29.33)
- Initial Treatment Period - Placebo: Initial Treatment Period - Placebo (n=94, PYE=27.93)
- Maintenance Treatment Period - Tralokinumab 300 Q2W: Maintenance Treatment Period - Tralokinumab 300 Q2W (n=11, PYE=5.61)
- Maintenance Treatment Period - Tralokinumab 300 Q4W: Maintenance Treatment Period - Tralokinumab 300 Q4W (n=13, PYE=6.78)
- Maintenance Treatment Period - Tralokinumab 150 Q2W: Maintenance Treatment Period - Tralokinumab 150 Q2W (n=12, PYE=6.40)
- Maintenance Treatment Period - Tralokinumab 150 Q4W: Maintenance Treatment Period - Tralokinumab 150 Q4W (n=14, PYE=6.53)
- Maintenance Treatment Period - Placebo: Maintenance Treatment Period - Placebo (n=6, PYE=2.98)
- Open-label Treatment - Tralokinumab 300 Q2W + Optional TCS: Open-label Treatment - Tralokinumab 300 Q2W + optional TCS (n=234, PYE=151.12)
- Safety Follow-up: Safety Follow-up (n=234, PYE=54.00)
Arm/Group | Initial Treatment Period - Tralokinumab 300 Q2W | Initial Treatment Period - Tralokinumab 150 Q2W | Initial Treatment Period - Placebo | Maintenance Treatment Period - Tralokinumab 300 Q2W | Maintenance Treatment Period - Tralokinumab 300 Q4W | Maintenance Treatment Period - Tralokinumab 150 Q2W | Maintenance Treatment Period - Tralokinumab 150 Q4W | Maintenance Treatment Period - Placebo | Open-label Treatment - Tralokinumab 300 Q2W + Optional TCS | Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/98 | 0/94 | 0/11 | 0/13 | 0/12 | 0/14 | 0/6 | 0/234 | 0/234
Serious Adverse Events (participants affected / at risk) | 1/97 | 3/98 | 5/94 | 0/11 | 0/13 | 0/12 | 0/14 | 0/6 | 7/234 | 3/234
Other Adverse Events (participants affected / at risk) | 44/97 | 47/98 | 36/94 | 7/11 | 6/13 | 7/12 | 8/14 | 4/6 | 100/234 | 16/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period - Tralokinumab 300 Q2W (N=97) | Initial Treatment Period - Tralokinumab 150 Q2W (N=98) | Initial Treatment Period - Placebo (N=94) | Maintenance Treatment Period - Tralokinumab 300 Q2W (N=11) | Maintenance Treatment Period - Tralokinumab 300 Q4W (N=13) | Maintenance Treatment Period - Tralokinumab 150 Q2W (N=12) | Maintenance Treatment Period - Tralokinumab 150 Q4W (N=14) | Maintenance Treatment Period - Placebo (N=6) | Open-label Treatment - Tralokinumab 300 Q2W + Optional TCS (N=234) | Safety Follow-up (N=234)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia nervosa (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obsessive-compulsive disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Treatment Period - Tralokinumab 300 Q2W (N=97) | Initial Treatment Period - Tralokinumab 150 Q2W (N=98) | Initial Treatment Period - Placebo (N=94) | Maintenance Treatment Period - Tralokinumab 300 Q2W (N=11) | Maintenance Treatment Period - Tralokinumab 300 Q4W (N=13) | Maintenance Treatment Period - Tralokinumab 150 Q2W (N=12) | Maintenance Treatment Period - Tralokinumab 150 Q4W (N=14) | Maintenance Treatment Period - Placebo (N=6) | Open-label Treatment - Tralokinumab 300 Q2W + Optional TCS (N=234) | Safety Follow-up (N=234)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 2 (3) | 6 (9) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 10 (16) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 2 (12) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 2 (2)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 11 (11) | 8 (10) | 4 (5) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 25 (34) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 12 (16) | 19 (22) | 8 (10) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 44 (60) | 1 (2)
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (17) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 (7) | 12 (16) | 11 (15) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 19 (26) | 8 (9)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 18 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-centre publication within 18 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (2):
  • Study Protocol (2020-02-06): https://cdn.clinicaltrials.gov/large-docs/61/NCT03526861/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT03526861/SAP_001.pdf